CLINICAL TRIAL: NCT02458768
Title: A Multicenter, Randomized, Open Label, Parallel Study to Evaluate the Efficacy & Safety of s.c. Administration of IVF-M HP Inj. Versus Menopur® Inj. in Infertility Women Undergoing Controlled Ovarian Hyperstimulation for Assisted Reproductive Technologies (ART) Such as in Vitro Fertilization-embryo Transfer (IVF-ET)
Brief Title: Multicenter, Randomized, Open Label, Parallel Study to Evaluate the Efficacy & Safety of IVF-M HP Inj. vs. Menopur® Inj.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-IMHCL001
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

ARMS (2):
- IVF-M HP Inj. (Experimental): administration was initiated on the mean menstrual cycle day (MCD) 2 or 3 and made by subcutaneous injection.
  Although the recommended initial dose of Investigational Product (IP) was 225 IU, adjustment was allowed according to the patient's individual response based on the monitoring (blood estradiol (E2) concentration and ultrasonography results).
  Interventions: Drug: IVF-M HP Inj.
- Menopur® Inj. (Active Comparator): administration was initiated on the mean menstrual cycle day (MCD) 2 or 3 and made by subcutaneous injection.
  Although the recommended initial dose of Investigational Product (IP) was 225 IU, adjustment was allowed according to the patient's individual response based on the monitoring (blood estradiol (E2) concentration and ultrasonography results).
  Interventions: Drug: Menopur® Inj.

INTERVENTIONS:
Drug: IVF-M HP Inj.
  Arms: IVF-M HP Inj.
Drug: Menopur® Inj.
  Arms: Menopur® Inj.

SUMMARY:
The objective of this study was to demonstrate the non-inferiority of IVFM HP Inj. by evaluating its efficacy versus Menopur® Inj. in infertility women undergoing the in vitro fertilization and embryo transfer (IVF-ET) among the assisted reproductive technologies.

ELIGIBILITY:
Inclusion Criteria:

* Adult women from 20 through 39 years of age at the screening
* Subjects with the mean menstrual cycle day (MCD) of 25 to 35 days
* Subjects with the Follicle Stimulating Hormone (FSH) concentration at the screening not exceeding the upper limit of the normal range (ULN)
* Those diagnosed with infertility due to at least one of the following causes of infertility

  * Fallopian tubal factor
  * Infertility due to unknown cause
  * Male infertility
  * Complex factor
* Subjects with the normal ovarian and uterine function
* Subjects with not more than 3 times of the prior experience of in vitro fertilization
* Subjects who had neither administered clomiphene citrate within 30 days nor gonadotropin within 14 days of the IP administration day
* Subjects who were informed on the objective, method and effect etc. of the clinical study and signed the informed consent form

Exclusion Criteria:

* Subjects contraindicated to pregnancy
* Subjects with BMI > 30 (BMI; kg/m2)
* Subjects diagnosed with polycystic ovary syndrome (PCOS)
* Subjects who had experienced previously at least Grade 4 ovarian hyperstimulation syndrome (OHSS)
* Subjects with poor response to gonadotropin (According to the Bologna criteria* below) *At least two of the following three features must be present:

  ① Advanced maternal age (>=40 years) or any other risk factor for Poor Ovarian Response (POR)

  ② A previous POR (<=3 oocyte with a conventional stimulation protocol)

  ③ An abnormal ovarian reserve test (i.e. Antral follicle Count (AFC) < 5 follicles or Anti-Mullerian hormone (AMH) < 0.5 ng/ml)
* Those with abnormal metrorrhagia due to unknown cause at the screening
* Subjects with submucosal uterine leiomyoma
* Subjects with at least borderline ovarian tumor
* Subjects with a history or malignant tumor in breast
* Subjects with hydrosalpinx not removed by operation
* Subjects with the Thyroid Stimulating Hormone (TSH) level out of the normal range at the screening
* Subjects with a history of malignant tumor within 5 years prior to the screening
* Subjects with severe disease potentially affecting the study such as pituitary insufficiency upon the investigator's judgment (e.g., heart failure, renal failure, hepatic failure or adrenal insufficiency etc.)
* Subject with HIV- or syphilis-positive result at the screening
* Subjects with a psychiatric disorder at the screening or those who failed in understanding the objective and method of this clinical study
* Subject diagnosed with alcohol or drug abuse within 3 months prior to the screening
* Subjects with a history of hypersensitivity to the investigational products of this clinical study
* Subjects with a current or history of thromboembolism in vein or artery
* Subjects with a history of genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
* Subjects who had participated in another clinical study related to a drug administration after the enrollment in this study or who had participated in another clinical study within 3 months prior to the enrollment in this study
* Others including the subjects for whom it was considered difficult to conduct this clinical study upon the principal investigator's judgment

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- IVF-M HP Inj.: Administration was initiated on the mean menstrual cycle day (MCD) 2 or 3 and made by subcutaneous injection.
  Although the recommended initial dose of Investigational Product (IP) was 225 IU, adjustment was allowed according to the patient's individual response based on the monitoring (blood estradiol (E2) concentration and ultrasonography results).
  IVF-M HP Inj.
- Menopur® Inj.: Administration was initiated on the mean menstrual cycle day (MCD) 2 or 3 and made by subcutaneous injection.
  Although the recommended initial dose of Investigational Product (IP) was 225 IU, adjustment was allowed according to the patient's individual response based on the monitoring (blood estradiol (E2) concentration and ultrasonography results).
  Menopur® Inj.
Period: Overall Study
Arm/Group | IVF-M HP Inj. | Menopur® Inj.
Started | 57 | 55
Completed | 50 | 50
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: Per-Protocol Set
Groups:
- Total: Total of all reporting groups
Arm/Group | IVF-M HP Inj. | Menopur® Inj. | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.05 (3.09) | 33.39 (3.19) | 33.21 (3.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Retrieved Oocytes
Time Frame: 36 hrs (±3 hrs) after administration of the ovulation stimulant
Population: Per-Protocol Set
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | IVF-M HP Inj. | Menopur® Inj.
Number analyzed (Participants) | 44 | 41
Oocytes | 13.14 (7.62) | 10.29 (6.65)

ADVERSE EVENTS:
Description: Among the 112 subjects randomized in this clinical study, one subject did not receive Investigational Product in the Menopur® Inj. group. This subject did not included in the Safety set. So total 111 subjects were included in the Safety set.
Arm/Group | IVF-M HP Inj. | Menopur® Inj.
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/54
Other Adverse Events (participants affected / at risk) | 13/57 | 16/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IVF-M HP Inj. (N=57) | Menopur® Inj. (N=54)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IVF-M HP Inj. (N=57) | Menopur® Inj. (N=54)
Abdominal distension (Gastrointestinal disorders) | 2 | 6
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 5
Abdominal discomfort (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 1 | 4
Lethargy (General disorders) | 3 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No